CLINICAL TRIAL: NCT05451849
Title: A Phase 1/2 Single Arm Open-Label Clinical Trial of TC-510 In Patients With Advanced Mesothelin-Expressing Cancer
Brief Title: A Phase 1/2 Trial of TC-510 In Patients With Advanced Mesothelin-Expressing Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TCR2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCR2-21-01
Record Dates: First submitted 2022-06-21; First posted 2022-07-11 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Mesothelioma; Mesotheliomas Pleural; Mesothelioma, Malignant; Mesothelioma Peritoneum; Ovarian Cancer; Ovarian Serous Adenocarcinoma; Pancreatic Cancer; Pancreatic Adenocarcinoma; Colorectal Cancer; Triple Negative Breast Cancer; TNBC - Triple-Negative Breast Cancer; Ovarian Adenocarcinoma; Pancreatic Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Cholangiocarcinoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant; Ovarian Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Cholangiocarcinoma; Carcinoma, Non-Small-Cell Lung | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lymphodepletion followed by TC-510 (Experimental): Lymphodepletion (fludarabine and cyclophosphamide) followed by TC-510 T cells
  Interventions: Biological: TC-510; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TC-510 — TC-510
Drug: Fludarabine — Fludarabine
Drug: Cyclophosphamide — Cyclophosphamide

SUMMARY:
TC-510 is a novel cell therapy that consists of autologous genetically engineered T cells expressing two synthetic constructs: first, a single-domain antibody that recognizes human Mesothelin, fused to the CD3-epsilon subunit which, upon expression, is incorporated into the endogenous T cell receptor (TCR) complex and second, a PD-1:CD28 switch receptor, which is expressed on the surface of the T cell, independently from the TCR. The PD-1:CD28 switch receptor comprises the PD-1 extracellular domain fused to the CD28 intracellular domain via a transmembrane domain. Thus, the switch is designed to produce a costimulatory signal upon engagement with PD-L1 on cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age at the time the Informed Consent is signed.
* Patient has a pathologically confirmed diagnosis of either MPM, Serous Ovarian Adenocarcinoma, Pancreatic Adenocarcinoma, TNBC, and Colorectal Cancer
* Patient's tumor has been reviewed with confirmed positive MSLN expression on >/= 50% of tumor cells that are 1+, 2+ and/or 3+ by immunohistochemistry. Patients with epithelioid MPM, confirmation of MSLN expression is not required prior to enrollment.
* Prior to TC-510 infusion, patients must have received at least 1 but no more than 5 systemic therapies for metastatic or unresectable disease with more details provided in the protocol
* Patients has an ECOG performance status 0 or 1
* Patient is fit for leukapheresis and has adequate venous access for the cell collection.
* Patient must have adequate organ function as indicated by the laboratory values in the clinical protocol

Exclusion Criteria:

* Inability to follow the procedures of the study
* Known or suspected non-compliance, drug, or alcohol use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1 - Establish the recommended Phase 2 dose (RP2D) according to dose-limiting toxicity (DLT) of defined adverse events. | DLTs within 28 days post-treatment
  Phase 1 -The number and percent of patients in the DLT evaluable set who experienced DLTs from the first administration of study drug up to 28 days post study drug treatment will be summarized by dosing group
Phase 2 - Overall Response Rate (ORR) | Up to 2 years post-treatment
  ORR is defined as incidence of complete responses or partial responses as assessed by RECIST v1.1
Phase 2 - Disease Control Rate (DCR) | Up to 2 years post-treatment
  DCR defined as a composite of ORR and stable disease (SD) lasting at least 8 weeks.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - National Cancer Institute, Bethesda, Maryland
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - SCRI Oncology Partners, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided